CLINICAL TRIAL: NCT06635291
Title: Improving the Diagnostic Accuracy of Children with Disorders of Consciousness in the REhabilitation Process (IDeAl DesiRE)
Brief Title: Improving the Diagnostic Accuracy of Children with DoC (IDeAl DesiRE)
Acronym: IDeAl DesiRE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 1108
Record Dates: First submitted 2024-09-10; First posted 2024-10-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Acquired Brain Injury; Disorder of Consciousness
Keywords: brain injury; disorder of consciousness; diagnosis; behavioral scale; children; pediatric
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The present study aims to investigate the clinical evolution of children with severe ABI and DoC both by using the traditional behavioral scales, namely the CRS-R, CRS-P and CNCS, and by trying to establish whether it is possible to identify any clinical markers of Emergency (E-Markers). E-Markers are behaviors that indicate a content of consciousness irrespective of the processes investigated by behavioral scales, thus they could be combined with the items of these scales to improve the diagnosis.

A particular focus will be given to the identification of specific E-Markers for children aged less than 12 months, for which the CRS-P scale cannot be used. In this case, the E-markers will be compared with the specific developmental stages of newborns, giving great importance to motor abilities.

DETAILED DESCRIPTION:
The assessment of the state of consciousness (CS) after an Acquired Brain Injury (ABI) is a complex and challenging process because of the clinical complexity of patients suffering from this condition. The most widely used measure to assess disturbance of consciousness (DoC) is the Coma Recovery Scale Revised (CRS-R), which is considered the gold standard for bedside assessments. This scale, even though validated for the adult population, has been recommended also for the pediatric population, considering the absence of tools designed to address children. In 2019, to fill this gap, Slomine and collaborators developed a pediatric form of the CRS, namely the Coma Recovery Scale for Pediatrics (CRS-P), but, up to now, it has been exclusively tested in typically developing children. Another tool frequently used to assess the DoC, even in pediatric age, is the Rappaport Coma Near Coma Scale (CNCS). In a recent study of our group, a statistically significant agreement between the CRS-R and the CNCS was found; however, the CNCS was found to better define patients' status in the emergency phase from minimally conscious state, while the CRS-R demonstrated to have lower DoC scoring ability in the presence of severe motor impairment. These results suggest new challenges for the diagnostic process, considering that the risk of misdiagnosis is still high.

The present study aims to investigate the clinical evolution of children with severe ABI and DoC both by using the traditional behavioral scales, namely the CRS-R, CRS-P and CNCS, and by trying to establish whether it is possible to identify any clinical markers of Emergency (E-Markers). E-Markers are behaviors that indicate a content of consciousness irrespective of the processes investigated by behavioral scales, thus they could be combined with the items of these scales to improve the diagnosis.

A particular focus will be given to the identification of specific E-Markers for children aged less than 12 months, for which the CRS-P scale cannot be used. In this case, the E-markers will be compared with the specific developmental stages of newborns, giving great importance to motor abilities; for this subgroup of children a small sample size is expected, which could not allow obtaining precise statistical data; however, results could lead to draw some relevant preliminary considerations.

For the whole sample, the effects of the various clinical, demographic and personal variables will be evaluated on functional outcome, intended as level of consciousness, disability degree and recovery level. Data based on neurophysiological and/or neuroimaging data will also be considered.

The investigators hypothesize that E-Markers may help clinicians to evaluate patients' clinical evolution earlier than behavioral scales.

ELIGIBILITY:
Inclusion Criteria:

* suffering from an ABI due to: traumatic brain injury, hypoxic events/anoxia, cerebral infections, cerebrovascular accident;
* age: 2 months-25.11 years;
* having a Glasgow Coma Scale (GCS; Teasdale & Jennett, 1974) at injury or onset ≤8);
* being in vegetative state (VS) or minimally conscious state (MCS) at admission;
* being in subacute or chronic phase.

Exclusion Criteria:

- ABI due to brain tumor or neurodegenerative disease.

Ages: 2 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population is composed of children and young adults suffering from an ABI admitted in the research timeframe to Scientifc Institute, IRCCS E. Medea, Bosisio Parini, Lecco, Italy.
  A total of 113 patients is required for the study. The calculation of the sample size was based on the comparison of the diagnostic capacity of the CRS-R with addition of E-markers and CRS-R without the addition of E-markers. This comparison has been analyzed using the area under the ROC curve. Assuming a percentage of patients emerging from a disorder of consciousness within the first 3 months after the ABI of 40% and an AUC of the CRS-R scale without the addition of E-markers of 0.7 (internal historical data), to identify a difference in the AUC of 0.15, with a power of 80% and a type I error of 5%, it is necessary to enroll 113 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) | CRS-R is administered at the time of admission (T0) and at 2 months (T1), 3 months (T3) and 6 months after the event (T4).
  The CRS-R is a behavioral scale used to assess level of consciousness in patients with disorders of consciousness. It consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level.
Rappaport Coma/Near Coma Scale (CNCS) | CNCS is administered at the time of admission (T0) and at 2 months (T1), 3 months (T3) and 6 months after the event (T4).
  The Rappaport Coma/Near Coma Scale is a behavioral scale designed to assess neurobehavioral status among patients who have sustained a severe brain injury, being in vegetative or near-vegetative state. It is composed of 11 items, assessing dysfunction in the sensory and perceptual domains, and describes the severity of primitive response deficits. Each item is scored on a 3-point rating scale (0, 2, and 4), with lower scores indicating better neurobehavioral functioning. A final level of Awareness/Responsivity is provided, ranging from 0 to 5, with lower scores indicating lower functioning.
Coma Recovery Scale for Pediatrics (CRS-P) | CRS-P is administered at the time of admission (T0) and at 2 months (T1), 3 months (T3) and 6 months after the event (T4).
  The CRS-P is a modified version of the Coma Recovery Scale-Revised (CRS-R), developed by Slomine and colleagues in 2019 to better evaluate the population of children with disorders of consciousness compared to the original scale, which was designed for the adults. It consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level, as for the CRS-R. Modifications include stimuli used, administration guidelines and scoring criteria. The overall score ranges from 0 to 23. Lower scores indicate worse functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute, IRCCS E. Medea, Bosisio Parini, Lecco, Italy

REFERENCES:
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Practice guideline update recommendations summary: Disorders of consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Neurology. 2018 Sep 4;91(10):450-460. doi: 10.1212/WNL.0000000000005926. Epub 2018 Aug 8. PMID 30089618
- [Background] Slomine BS, Suskauer SJ, Nicholson R, Giacino JT. Preliminary validation of the coma recovery scale for pediatrics in typically developing young children. Brain Inj. 2019;33(13-14):1640-1645. doi: 10.1080/02699052.2019.1658221. Epub 2019 Aug 28. PMID 31462082
- [Background] Frigerio S, Molteni E, Colombo K, Pastore V, Fedeli C, Galbiati S, Strazzer S. Neuropsychological assessment through Coma Recovery Scale-Revised and Coma/Near Coma Scale in a sample of pediatric patients with disorder of consciousness. J Neurol. 2023 Feb;270(2):1019-1029. doi: 10.1007/s00415-022-11456-6. Epub 2022 Nov 5. PMID 36335241